CLINICAL TRIAL: NCT02214043
Title: Clinical Characteristics of Acute Pulmonary Embolism in Chinese Population
Status: Completed | Type: Observational
Sponsor: Chinese Pulmonary Vascular Disease Research Group (Other)
Responsible Party: Sponsor
Other Study IDs: APEINCP
Record Dates: First submitted 2014-02-03; First posted 2014-08-12 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2016-07

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — BNP，D-dimer
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group 2
- group 1

SUMMARY:
There are no special clinical characteristics of acute pulmonary embolism in Chinese population.

ELIGIBILITY:
Inclusion Criteria:

* the symptomatic acute PE confirmed by objective examination

Exclusion Criteria:

* congestive heart failure
* chronic obstructive pulmonary disease;
* a prior documented episode of PE or DVT
* renal dysfunction;
* a life expectancy of less than 6 months

Ages: 15 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Acute pulmonary embolism in Chinese population
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2012-01; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
The primary end point of the present study was symptomatic, objectively confirmed recurrent fatal or nonfatal VTE. | 60 months

SECONDARY OUTCOMES:
The second end point was death (all cause death and PE-related death). | 60 months
  If the participant died, the relatives need provided the written medical record on the death.

CONTACTS AND LOCATIONS:
Overall Officials: Zhihong Liu, Doctor, Study Chair — Chinese pulmonary vascular disease organization group
Locations (1):
- Center of pumonary vascular diseases, Beijing, China